CLINICAL TRIAL: NCT06344052
Title: A Phase 2 Study to Assess the Efficacy of SP-002 with Vismodegib for the Treatment of Locally Advanced Basal Cell Carcinoma
Brief Title: To Assess the Safety and Efficacy of SP-002 with Vismodegib for the Treatment of Locally Advanced Basal Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stamford Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP-002-004
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Basal Cell Carcinoma
Keywords: locally advanced
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): vismodegib, with 3 cycles SP-002
  Interventions: Drug: SP-002; Drug: Vismodegib
- Arm 2 (Experimental): vismodegib, with 1 cycles SP-002
  Interventions: Drug: SP-002; Drug: Vismodegib
- Arm 3 (Placebo Comparator): vismodegib monotherapy
  Interventions: Drug: Vismodegib

INTERVENTIONS:
Drug: SP-002 — SP-002 is a replication deficient adenovirus-5 encoding human interferon gamma (IFNγ), designed for intra-tumoral administration
  Arms: Arm 1; Arm 2
Drug: Vismodegib — The HHPI vismodegib is currently indicated for the treatment of adult patients with metastatic BCC, or with laBCC where surgery and/or radiation therapy are not appropriate.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of using SP-002 in participants with locally advanced Basal cell carcinoma. The main question it aims to answer is what the objective response rate for a basal cell carcinoma tumor is following 1 or 3 cycles of SP-002 treatment given as an add-on to hedgehog pathway inhibitor therapy.

Researchers will compare the objective response rate for treated Basal cell carcinoma tumors between 3 treatment Arms.

* Arm 1 participants will receive daily hedgehog pathway inhibitor, and 3 cycles of SP-002 treatment.
* Arm 2 participants will receive daily hedgehog pathway inhibitor, and 1 cycle of SP-002 treatment.
* Arm 3 participants will receive daily hedgehog pathway inhibitor only.

DETAILED DESCRIPTION:
This is a Phase 2, 3-arm, multi-center, open-label, randomized, clinical study to evaluate the efficacy of SP-002 in combination with vismodegib in subjects with locally advanced Basal cell carcinoma.

The study will be completed in 2 consecutive parts. Each part consists of a screening period, a treatment period, and a follow-up period.

* Part A: 20 participants who meet study entry criteria will be randomized in a 1:1 ratio into 2 treatment arms (Arm 2 and Arm 3) and will provide preliminary safety and performance in a population with target Basal cell carcinoma lesions.
* Part B: 60 participants who meet study entry criteria will be randomized in a 1:1:1 ratio into 3 treatment arms (Arm 1, Arm 2, and Arm 3) in a population with target Basal cell carcinoma lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent prior to initiation of study-specified procedures.
2. Subject is 18 years of age or older.
3. Eastern Cooperative Oncology Group performance status 0, 1 or 2.
4. Subject has a single lesion that is histologically confirmed as BCC. The externally visible component of the lesions should be at least 1 cm in one dimension to facilitate accurate and reproducible measurement, to 5 cm at longest diameter, that in the opinion of the investigator:

   A. is considered not a good candidate for surgery or has recurred after definitive surgical treatment and curative surgical resection is unlikely. OR

   B. subject has a medical contraindication to surgery where acceptable medical contraindications to surgery include:
   * Anticipated substantial morbidity and/or deformity from surgery (e.g., removal of all or part of a vital facial structure, such as nose, ear, eyelid, eye; or requirement for limb amputation).
   * Medical conditions predisposing to poor surgical outcome (e.g., diabetes with history of poor wound healing).
   * Other conditions considered to be medically contraindicating must be discussed with the Medical Monitor before enrolling the subject.

   A copy of the surgical consultation note must be provided. laBCC with prior history of or ongoing HPPI treatment are eligible under the following conditions:
   * Achieved objective response with disease progression >3 months after treatment discontinuation.
   * Achieve best response of PR with persistent disease that continues to meet study inclusion criteria and has been off treatment for at least 3 months.

   Note: where the subject has >1 lesion, one lesion may be selected for treatment at the discretion of the investigator.
5. Radiotherapy is contraindicated or inappropriate in the opinion of the investigator, for example, hypersensitivity to radiation due to genetic syndrome such as Gorlin syndrome, limitations because of location of tumor, or anticipated significant morbidity, loss of function, or unacceptable cosmetic outcomes. Patients with Basal Cell Nevus Syndrome (Gorlin syndrome) may enroll in this study but must meet the criteria for locally advanced or listed above.
6. Subject is able and willing to comply with all study requirements including biopsies at baseline and during the study. Biopsy 3-4 mm preferred, biopsies must be <25% of the area the tumor. Screening biopsies performed 1-12 weeks before Day 1.
7. Subject has adequate hematopoietic capacity, as defined by the following:

   * Neutrophil count >1,500/mm3
   * Hemoglobin >9 g/dL
   * Platelet count >100,000/ mm3
   * Prothrombin international normalized ratio <1.5
8. Subject has adequate hepatic function, as defined by the following:

   * Total bilirubin <1.5 × the upper limit of normal (ULN) or within 3 × the ULN for patients with Gilbert disease
   * Aspartate aminotransferase, alanine aminotransferase or alkaline phosphate <2 × the ULN
9. Adequate renal function, as defined by the following:

   * Creatinine <1.5 x ULN
10. For female subjects of childbearing potential*, agreement to use two acceptable methods of contraception (including one barrier method), during the study and for at least (per United States Prescribing Information [USPI]) 24 months after discontinuation of vismodegib.

    For male subjects with female partners of childbearing potential*, agreement to use a latex condom, and to advise their female partner to use an additional method of contraception during the study and for at least (per USPI) 24 months after discontinuation of vismodegib.
11. Subjects agree not to donate blood or blood products during the study and for at least (per USPI) 24 months after discontinuation of vismodegib; male subjects agree not to donate sperm during the study and for at least 2 months after discontinuation of vismodegib.

    * Childbearing potential is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in the absence of other biological causes. In addition, females under the age of 55 years must have a documented serum follicle stimulating hormone level >40 mIU/mL to confirm menopause.

Exclusion Criteria:

1. laBCC that has progressed on systemic HHPI therapy as defined below:

   * Best response of progressive disease (primary progression).
   * Objective response followed by disease progression while on HHPI treatment.
   * laBCC with a best response of stable disease on systemic HHPI treatment.
2. laBCC that has recurred in the same location after two or more surgical procedures, or that has recurred following radiation therapy.
3. laBCC that has bone involvement (radiologically confirmed if clinically suspected).
4. laBCC with invasion of underlying soft tissue that is not accessible by standard syringe/needle.
5. Patients with evidence of metastatic BCC.
6. Female subjects who are lactating or pregnant.
7. Life expectancy of <12 weeks.
8. Concurrent non-protocol-specified anti-tumor therapy (e.g., chemotherapy, other targeted therapy, or radiation therapy).
9. Recent (within 4 weeks of Day 1), current, or planned participation in an experimental drug study.
10. History of other malignancies within 3 years of Day 1, except for tumors with a negligible risk for metastasis or death, such as adequately treated basal and squamous-cell carcinoma of the skin, ductal carcinoma in situ of the breast, or carcinoma in situ of the cervix.
11. Uncontrolled medical illnesses such as infection requiring treatment with intravenous antibiotics.
12. History of other stable disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or renders the subject at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Week 26
  ORR defined as the proportion of subjects who achieve complete response (CR) or partial response (PR) of the target lesion based on central review at any time point.

SECONDARY OUTCOMES:
Duration of response | Month 36
  DOR defined as the time interval between the date of first response (CR or PR) of the target lesion to the date of disease progression or death from any cause. Disease progression as assessed by central review.
Progressive free survival | Month 36
  PFS defined as the time interval between the date of randomization/start of treatment to the date of first documented progression of the target tumor or death. If a subject has not had an event, PFS is censored at the date of last adequate tumor assessment. Rate of disease progression of the target tumor as assessed by central review.
Overall survival (OS) | Month 36
  OS defined as the time interval between the date of randomization and the date of death. If a subject has not had an event, the patient will be censored at the date of the last study visit attended.
Objective Response Rate (ORR) / Complete Response (CR) / Partial Response (PR) | Month 36
  ORR/CR/PR by investigator assessment (color photography/imaging [RECIST-measurable]).
Number of subjects discontinuing treatment with SP-002 and/or vismodegib due to toxicity. | Month 36
  Safety of Participants
Number of subjects with delays to SP-002 and/or vismodegib dosing due to toxicity. | Month 36
  Safety of Participants
Incidence and severity of SP-002 and/or vismodegib related AEs. | Month 36
  Safety of Participants

CONTACTS AND LOCATIONS:
Overall Officials: Stamford Pharmaceuticals, Study Chair — Stamford Pharmaceuticals
Locations (10):
- United States (10):
  - Research Site, Phoenix, Arizona
  - Research Site, Boca Raton, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Cutler Bay, Florida
  - Research Site, Rockville, Maryland
  - Research Site, Lee's Summit, Missouri
  - Research Site, Rochester, New York
  - Research Site, Cedar Park, Texas
  - Research Site, Humble, Texas
  - Research Site, Longview, Texas

IPD SHARING:
Plan to Share IPD: No